CLINICAL TRIAL: NCT04796935
Title: An Open-Label, Parallel, Randomized Study to Evaluate the Performance of Needle Placements for Diagnostic and Therapeutic Neuraxial Procedures, Using a Handheld Tactile Imaging-based Method Versus Palpation
Brief Title: A Study to Test Performance of Needle Placements for Neuraxial Procedures Using Tactile Imaging vs Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IntuiTap Medical, Inc (Industry)
Collaborators: ICON plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: INT-001
Record Dates: First submitted 2021-03-10; First posted 2021-03-15 (Actual); Results first posted 2024-06-06 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Central Nervous System Infections; Pseudotumor Cerebri; Neurological Disorder; Cancer; Obstetric Procedure Pain; Orthopedic Procedure Pain; Post-Dural Puncture Headache
Keywords: Diagnostic spinal puncture; Therapeutic spinal puncture; Lumbar puncture; Epidural; Neuraxial anesthesia; Blood patch; ESI
MeSH Terms: conditions — Central Nervous System Infections; Pseudotumor Cerebri; Nervous System Diseases; Neoplasms; Post-Dural Puncture Headache

STUDY DESIGN:
Intervention Model Description: An open-label, parallel, randomized study design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Experimental Group 1: Tactile Imaging (VerTouch) (Experimental): VerTouch used to identify and mark, or begin placement of a needle, at an insertion site.
  Interventions: Device: Tactile Imaging (VerTouch)
- Group 2: Control (palpation) (Active Comparator): Palpation used to identify and mark an insertion site.
  Interventions: Other: Control (palpation)

INTERVENTIONS:
Device: Tactile Imaging (VerTouch) — VerTouch device used to identify and mark, or begin placement of a needle at an insertion site. After the device is taken off the back, the procedure will continue in the usual manner.
  Arms: Experimental Group 1: Tactile Imaging (VerTouch)
Other: Control (palpation) — Control, palpation used to identify and mark an insertion site.
  Arms: Group 2: Control (palpation)

SUMMARY:
This study will compare the VerTouch device to the conventional palpation technique for performing diagnostic and therapeutic neuraxial procedures.

DETAILED DESCRIPTION:
Neuraxial procedures, in which a needle is inserted into the spinal canal through a gap in the vertebrae, are performed at a rate of nearly 13 million per year in the US, across a myriad of diagnostic and therapeutic clinical scenarios.

The standard of care involves manual palpation of the patient's back to detect the spinous processes (SPs) and estimate the location of the interspinous needle insertion site. While providers are trained to perform these procedures with meticulous precision and attention to detail, this technique remains highly inaccurate, often requiring multiple insertion attempts to properly place the needle. These attempts lead to patient pain and complications, such as traumatic taps and post-dural puncture (PDPH) headaches; unpredictable procedure times; and poor facility throughput.

The VerTouch device uses tactile imaging to offer a non-invasive, untethered, non radiation-producing solution for visualizing spinal anatomy in order to identify an ideal location for needle placement in a neuraxial procedure. The device can be used to mark the identified site with a surgical marker, or to begin placement of a needle or introducer at that site.

Study participants will be recruited in two parallel cohorts: the control (palpation) group or the tactile imaging (VerTouch) group, further stratified by procedure setting, including emergency medicine, neurology, and anesthesiology. Once an insertion site is marked with a marker or shallow placement of a needle or introducer, the procedure will continue in the usual manner for subjects in both groups.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 18 years and above, inclusive
2. Subjects scheduled for one of the following procedures:

   * Diagnostic LP (collection of CSF and/or measurement of ICP to diagnose hemorrhaging or neurological infections)
   * Therapeutic LP (intrathecal injection of therapeutic agents; drainage of CSF to treat pseudotumor cerebri)
   * Planned orthopedic or obstetric procedure, such as labor/induction, cesarean section, hysterectomy, or total hip/knee replacement, with neuraxial anesthesia (injection of anesthetic into spinal and/or epidural space to reduce pain during procedure)
   * Epidural blood patch (use of autologous blood to close holes in the dura mater and relieve PDPH)
3. Subjects having a BMI ≤42kg/m2

Exclusion Criteria:

1. Patient does not provide informed consent
2. Skin or soft tissue infection near the puncture site
3. Allergy to local anesthetic
4. Uncorrected coagulopathy
5. Acute spinal cord trauma
6. History of lumbar spinal surgery
7. Prior known failed neuraxial anesthesia
8. Diagnosed scoliosis, thoracic kyphosis, lumbar lordosis, scleroderma, or ankylosing spondylitis, or lumbar spinal stenosis
9. Incarcerated subjects

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2021-04-04 (Actual); Primary Completion 2021-11-24 (Actual); Study Completion 2021-11-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Health Science Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After enrollment, subjects meeting eligibility criteria were randomized; the rest were considered screen failures.
Period: Overall Study
Arm/Group | Experimental Group 1: Tactile Imaging (VerTouch) | Group 2: Control (Palpation)
Started | 42 | 48
Received Randomized Location Method | 30 | 46
Achieved Procedure Success (Procedure success was defined as confirmation of entry into the spinal canal using standard methods (e.g. return of cerebrospinal fluid from the needle).) | 30 | 41
Completed | 40 | 46
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Device not available | 1 | 0
Not completed — Trained provider not available | 1 | 0

BASELINE CHARACTERISTICS:
Population: This population includes all randomized subjects and is referred to as the Intent-to-Treat (ITT) population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Group 1: Tactile Imaging (VerTouch) | Group 2: Control (Palpation) | Total
Number analyzed (Participants) | 42 | 48 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Per-Protocol (PP) excludes subjects that did not receive the randomized method and/or achieve a procedure success.
  years
    ITT | 43.8 (17.67) | 40.5 (18.47) | 42.0 (18.07)
    PP: number analyzed (Participants) | 25 | 41 | 66
    PP | 41.4 (15.55) | 39.3 (17.78) | 40.1 (16.8)
Age, Customized [Count of Participants; unit: Participants] — Population: Per-Protocol (PP) excludes subjects that did not receive the randomized method and/or achieve a procedure success.
  Participants
    ITT: Adolescent (<22) | 2 | 3 | 5
    ITT: Young Adult (22-40) | 19 | 28 | 47
    ITT: Middle-aged Adult (41-65) | 15 | 10 | 25
    ITT: Older Adult (>65) | 6 | 7 | 13
    PP: number analyzed (Participants) | 25 | 41 | 66
    PP: Adolescent (<22) | 1 | 3 | 4
    PP: Young Adult (22-40) | 12 | 25 | 37
    PP: Middle-aged Adult (41-65) | 10 | 8 | 18
    PP: Older Adult (>65) | 2 | 5 | 7
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Per-Protocol (PP) excludes subjects that did not receive the randomized method and/or achieve a procedure success.
  Participants
    ITT: Female | 29 | 36 | 65
    ITT: Male | 13 | 12 | 25
    PP: number analyzed (Participants) | 25 | 41 | 66
    PP: Female | 21 | 32 | 53
    PP: Male | 4 | 9 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Per-Protocol (PP) excludes subjects that did not receive the randomized method and/or achieve a procedure success.
  Participants
    ITT: Hispanic or Latino | 9 | 14 | 23
    ITT: Not Hispanic or Latino | 33 | 33 | 66
    ITT: Unknown or Not Reported | 0 | 1 | 1
    PP: number analyzed (Participants) | 25 | 41 | 66
    PP: Hispanic or Latino | 6 | 12 | 18
    PP: Not Hispanic or Latino | 19 | 28 | 47
    PP: Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Per-Protocol (PP) excludes subjects that did not receive the randomized method and/or achieve a procedure success.
  Participants
    ITT: American Indian or Alaska Native | 0 | 0 | 0
    ITT: Asian | 2 | 1 | 3
    ITT: Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
    ITT: Black or African American | 8 | 10 | 18
    ITT: White | 27 | 32 | 59
    ITT: More than one race | 0 | 0 | 0
    ITT: Unknown or Not Reported | 4 | 4 | 8
    PP: number analyzed (Participants) | 25 | 41 | 66
    PP: American Indian or Alaska Native | 0 | 0 | 0
    PP: Asian | 1 | 1 | 2
    PP: Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
    PP: Black or African American | 6 | 7 | 13
    PP: White | 16 | 29 | 45
    PP: More than one race | 0 | 0 | 0
    PP: Unknown or Not Reported | 1 | 3 | 4
Height [Mean (Standard Deviation); unit: cm] — Population: BMI could not be calculated for one ITT subject whose height was not recorded. Per-Protocol (PP) excludes subjects that did not receive the randomized method and/or achieve a procedure success.
  cm
    ITT: number analyzed (Participants) | 42 | 47 | 89
    ITT | 165.7 (9.53) | 165.3 (10.36) | 165.5 (9.93)
    PP: number analyzed (Participants) | 25 | 41 | 66
    PP | 163.5 (8.74) | 164.8 (10.45) | 164.3 (9.79)
Weight [Mean (Standard Deviation); unit: kg] — Population: Per-Protocol (PP) excludes subjects that did not receive the randomized method and/or achieve a procedure success.
  kg
    ITT | 81.6 (19.40) | 80.6 (17.71) | 81.0 (18.42)
    PP: number analyzed (Participants) | 25 | 41 | 66
    PP | 77.6 (18.44) | 79.9 (17.86) | 79.0 (17.97)
BMI [Mean (Standard Deviation); unit: kg/m^2] — BMI was calculated from subject height and weight, with units of kg/m^2. Population: BMI could not be calculated for one ITT subject whose height was not recorded. Per-Protocol (PP) excludes subjects that did not receive the randomized method and/or achieve a procedure success.
  kg/m^2
    ITT: number analyzed (Participants) | 42 | 47 | 89
    ITT | 29.6 (5.94) | 29.4 (6.56) | 29.5 (6.24)
    PP: number analyzed (Participants) | 25 | 41 | 66
    PP | 29.0 (6.10) | 29.5 (6.37) | 29.3 (6.37)
BMI, categorical [Count of Participants; unit: Participants] — Population: BMI could not be calculated for one ITT subject whose height was not recorded. Per-Protocol (PP) excludes subjects that did not receive the randomized method and/or achieve a procedure success.
  Participants
    ITT: number analyzed (Participants) | 42 | 47 | 89
    ITT: Underweight (<18.5) | 0 | 1 | 1
    ITT: Normal (18.5-24.9) | 10 | 15 | 25
    ITT: Overweight (25-29.9) | 11 | 9 | 20
    ITT: Class 1 Obesity (30-34.9) | 13 | 12 | 25
    ITT: Class 2-3 Obesity (≥35) | 8 | 10 | 18
    PP: number analyzed (Participants) | 25 | 41 | 66
    PP: Underweight (<18.5) | 0 | 1 | 1
    PP: Normal (18.5-24.9) | 6 | 12 | 18
    PP: Overweight (25-29.9) | 9 | 9 | 18
    PP: Class 1 Obesity (30-34.9) | 5 | 10 | 15
    PP: Class 2-3 Obesity (≥35) | 5 | 9 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Insertion Attempts
Description: Any forward movement of the needle following puncture of the skin, counted until confirmation of spinal canal access can be assessed.
Time Frame: End of procedure, 1 per participant
Population: Intent-to-Treat (ITT) includes all randomized subjects. Per-Protocol (PP) excludes subjects that did not receive the randomized method and/or achieve a procedure success. Number analyzed in each population refers to the subjects with data collected for the specific outcome measure.
Measure: Mean (Standard Deviation); unit: insertions
Arm/Group | Experimental Group 1: Tactile Imaging (VerTouch) | Group 2: Control (Palpation)
Number analyzed (Participants) | 42 | 48
insertions
  ITT: number analyzed (Participants) | 36 | 46
  ITT | 1.8 (0.26) | 2.2 (0.3)
  PP: number analyzed (Participants) | 25 | 41
  PP | 1.2 (0.66) | 2.1 (2.10)

2. Secondary Outcome: Incidence of First-insertion Success
Description: A case that does not require any reinsertions, but can include any number of redirections.
Time Frame: End of procedure, 1 per subject
Population: ITT includes all randomized subjects. PP excludes subjects that did not receive the randomized method and/or achieve a procedure success. Number analyzed in each population refers to the subjects with data recorded for the related outcome measure (insertions).
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Group 1: Tactile Imaging (VerTouch) | Group 2: Control (Palpation)
Number analyzed (Participants) | 42 | 48
Participants
  ITT: number analyzed (Participants) | 36 | 46
  ITT | 25 | 25
  PP: number analyzed (Participants) | 25 | 41
  PP | 21 | 25

3. Secondary Outcome: Number of Redirections
Description: Any forward movement of the needle in a new direction not preceded by withdrawal from the skin, counted until confirmation of spinal canal access can be assessed.
Time Frame: End of procedure, 1 per subject
Population: ITT includes all randomized subjects. PP excludes subjects that did not receive the randomized method and/or achieve a procedure success. Number analyzed in each population refers to the subjects with data collected for the specific outcome measure.
Measure: Mean (Standard Deviation); unit: redirections
Arm/Group | Experimental Group 1: Tactile Imaging (VerTouch) | Group 2: Control (Palpation)
Number analyzed (Participants) | 42 | 48
redirections
  ITT: number analyzed (Participants) | 37 | 46
  ITT | 4.5 (5.60) | 5.8 (8.44)
  PP: number analyzed (Participants) | 25 | 41
  PP | 2.5 (3.14) | 5.2 (8.31)

4. Secondary Outcome: Number of Passes
Description: Any forward movement of the needle, calculated as the sum of insertions and redirections.
Time Frame: End of procedure, 1 per subject
Population: ITT includes all randomized subjects. PP excludes subjects that did not receive the randomized method and/or achieve a procedure success. Number analyzed in each population refers to the subjects with data collected for the related outcome measures (insertions and redirections).
Measure: Mean (Standard Deviation); unit: passes
Arm/Group | Experimental Group 1: Tactile Imaging (VerTouch) | Group 2: Control (Palpation)
Number analyzed (Participants) | 42 | 48
passes
  ITT: number analyzed (Participants) | 36 | 46
  ITT | 6.4 (6.66) | 8.0 (9.78)
  PP: number analyzed (Participants) | 25 | 41
  PP | 3.8 (3.49) | 7.3 (9.62)

5. Secondary Outcome: Incidence of First-pass Success
Description: A case that does not require reinsertions or redirections.
Time Frame: End of procedure, 1 per subject
Population: ITT includes all randomized subjects. PP excludes subjects that did not receive the randomized method and/or achieve a procedure success. Number analyzed in each population refers to the subjects with data collected for the related outcome measures (insertions, redirections).
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Group 1: Tactile Imaging (VerTouch) | Group 2: Control (Palpation)
Number analyzed (Participants) | 42 | 48
Participants
  ITT: number analyzed (Participants) | 36 | 46
  ITT | 10 | 9
  PP: number analyzed (Participants) | 25 | 41
  PP | 9 | 9

6. Secondary Outcome: Subject Discomfort During Landmarking
Description: Evaluated using a 10-point Numeric Pain Rating Scale, where 1 is equivalent to no pain and 10 is equivalent to the worst possible pain.
Time Frame: End of procedure, 1 per subject
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Group 1: Tactile Imaging (VerTouch) | Group 2: Control (Palpation)
Number analyzed (Participants) | 42 | 48
score on a scale
  ITT: number analyzed (Participants) | 41 | 46
  ITT | 2.0 (2.17) | 1.9 (2.43)
  PP: number analyzed (Participants) | 25 | 41
  PP | 1.5 (1.66) | 1.5 (1.89)

7. Secondary Outcome: Provider Confidence With the Identified Insertion Site
Description: Evaluated using a 1-5 point Numeric Rating Scale where 1 is equivalent to not at all confident and 5 equivalent to completely confident.
Time Frame: End of procedure, 1 per subject
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Group 1: Tactile Imaging (VerTouch) | Group 2: Control (Palpation)
Number analyzed (Participants) | 40 | 46
score on a scale
  ITT | 3.6 (1.43) | 4.2 (0.97)
  PP: number analyzed (Participants) | 25 | 41
  PP | 4.0 (1.24) | 4.2 (0.97)

8. Other Pre Specified Outcome: Localization Time
Description: Time from first touch of draped patient to identification of an insertion site; for VerTouch, this is the time from VerTouch device placement to movement of the applicator to the identified insertion site.
Time Frame: End of procedure, 1 per subject
Population: PP excludes subjects that did not receive the randomized method and/or achieve a procedure success.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Experimental Group 1: Tactile Imaging (VerTouch) | Group 2: Control (Palpation)
Number analyzed (Participants) | 25 | 41
seconds | 197.3 (247.03) | 170.3 (300.12)

9. Other Pre Specified Outcome: Insertion Time
Description: Time from retrieval of marker or local-anesthetic assembly until no further needle advancements are made.
Time Frame: End of procedure, 1 per subject
Population: PP excludes subjects that did not receive the randomized method and/or achieve a procedure success.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Experimental Group 1: Tactile Imaging (VerTouch) | Group 2: Control (Palpation)
Number analyzed (Participants) | 25 | 41
seconds | 303.5 (600.79) | 301.8 (390.73)

10. Other Pre Specified Outcome: Total Procedure Time
Description: From positioning of the patient to removal of the drape from the subject's back.
Time Frame: End of procedure, 1 per subject
Population: PP excludes subjects that did not receive the randomized method and/or achieve a procedure success.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Experimental Group 1: Tactile Imaging (VerTouch) | Group 2: Control (Palpation)
Number analyzed (Participants) | 25 | 41
minutes | 19.3 (16.43) | 20.5 (28.03)

11. Other Pre Specified Outcome: Bone Contacts
Description: Number of times the needle contacts bone, counted until confirmation of spinal canal access can be assessed.
Time Frame: End of procedure, 1 per subject
Population: PP excludes subjects that did not receive the randomized method and/or achieve a procedure success.
Measure: Mean (Standard Deviation); unit: contacts
Arm/Group | Experimental Group 1: Tactile Imaging (VerTouch) | Group 2: Control (Palpation)
Number analyzed (Participants) | 25 | 41
contacts | 2.0 (6.04) | 2.9 (4.81)

12. Other Pre Specified Outcome: Incidence of Unintended Dural Puncture
Description: A case that results in puncture of the dura when it is not intended (i.e., in an epidural procedure).
Time Frame: End of procedure, 1 per subject
Population: All randomized subjects with data for the safety endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Group 1: Tactile Imaging (VerTouch) | Group 2: Control (Palpation)
Number analyzed (Participants) | 40 | 45
Participants | 0 | 0

13. Other Pre Specified Outcome: Incidence of Paresthesia During Needle Insertion
Description: A case in which paresthesia is experienced during needle insertion.
Time Frame: End of procedure, 1 per subject
Population: All randomized subjects with data for the safety endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Group 1: Tactile Imaging (VerTouch) | Group 2: Control (Palpation)
Number analyzed (Participants) | 40 | 45
Participants | 8 | 9

14. Other Pre Specified Outcome: Incidence of Traumatic Tap
Description: A case that results in visible blood aspiration.
Time Frame: End of procedure, 1 per subject
Population: All randomized subjects with data for the safety endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Group 1: Tactile Imaging (VerTouch) | Group 2: Control (Palpation)
Number analyzed (Participants) | 40 | 45
Participants | 1 | 4

15. Other Pre Specified Outcome: Incidence of Referral to Radiology
Description: A case in which the provider cannot perform the procedure at the bedside and refers the subject to radiology for the procedure to be completed under fluoroscopic guidance.
Time Frame: End of procedure, 1 per subject
Population: All randomized subjects with data for the safety endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Group 1: Tactile Imaging (VerTouch) | Group 2: Control (Palpation)
Number analyzed (Participants) | 40 | 45
Participants | 4 | 2

16. Other Pre Specified Outcome: Incidence of Conversion From Spinal to Epidural
Description: A case that the provider opts to complete using epidural anesthesia instead of spinal anesthesia.
Time Frame: End of procedure, 1 per subject
Population: All randomized subjects with data for the safety endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Group 1: Tactile Imaging (VerTouch) | Group 2: Control (Palpation)
Number analyzed (Participants) | 40 | 45
Participants | 0 | 0

17. Other Pre Specified Outcome: Incidence of Post-dural Puncture Headache
Description: A case that results in the patient experiencing one or more headache of any level of severity after the procedure and/or at follow-up.
Time Frame: Follow up, 3±2 days after procedure, 1 per subject
Population: All randomized subjects with data for the safety endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Group 1: Tactile Imaging (VerTouch) | Group 2: Control (Palpation)
Number analyzed (Participants) | 40 | 46
Participants | 9 | 16

ADVERSE EVENTS:
Time Frame: 3±2 days
Arm/Group | Experimental Group 1: Tactile Imaging (VerTouch) | Group 2: Control (Palpation)
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/48
Other Adverse Events (participants affected / at risk) | 2/42 | 1/48
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Group 1: Tactile Imaging (VerTouch) (N=42) | Group 2: Control (Palpation) (N=48)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) — VerTouch Group: determined unlikely to be related to device
Hemorrhage (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — VerTouch Group: determined unrelated to device
Back and Shoulder Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Palpation Arm: may have been related to study procedure but not study device (control group)

LIMITATIONS AND CAVEATS:
The enrollment period (April 2021-November 2021) was closed due to COVID concerns prior to reaching 96 evaluable subjects. Due to limitations in the emergency medicine setting at one site, emergency medicine providers at that site performed procedures for approximately half of the subjects enrolled in that site's neurology setting. Due to scheduling limitations, only MDs (including residents) performed procedures, and not all providers had the opportunity to use the device more than once.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-11-25): https://cdn.clinicaltrials.gov/large-docs/35/NCT04796935/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-22): https://cdn.clinicaltrials.gov/large-docs/35/NCT04796935/SAP_001.pdf